CLINICAL TRIAL: NCT02117128
Title: The Efficacy and Safety of Using Tranexamic Acid by Different Means to Reduce Blood Loss During Total Knee Replacement: a Randomized, Double-blind, Controlled Trial
Brief Title: The Efficacy and Safety of Using Tranexamic Acid by Different Means to Reduce Blood Loss During Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chenxiaoyong, Doctor-in-charge, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJODCT2014001
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Blood Loss
Keywords: Tranexamic Acid; Antifibrinolytic; Blood transfusion; Total knee arthroplasty
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tranexamic acid, IA group (Experimental): Tranexamic acid 1g, intra-articular injection, post-operationally
  Interventions: Drug: Tranexamic acid
- Tranexamic acid, IV group (Active Comparator): Tranexamic acid, 1g, intravenous injection, post-operationally
  Interventions: Drug: Tranexamic acid
- Tranexamic acid, IV+IA group (Experimental): Tranexamic acid, 1g, intravenous injection, post-operationally; Tranexamic acid, 1g, intra-articular injection, post-operationally
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid

SUMMARY:
We will investigate the efficacy and safety of using tranexamic acid by intravenous, intra-articular and combinational administration to reduce blood loss during total knee replacement. We hypothesize a combined intra-articular and single intravenous dose protocol of tranexamic acid may achieve a higher therapeutic concentration at the intra-articular and extra-articular bleeding site with little or no systemic absorption and subsequent systemic side effects.

DETAILED DESCRIPTION:
A randomized, double-blind, single-center, controlled and parallel-assigned study comparing the efficacy and safety of intravenous, intra-articular and combinational administration of tranexamic acid to reduce blood loss during total knee replacement. Subjects will be monitored for occurrence of any complications, particularly deep venous thrombosis and thromboembolism during the hospital stay and for 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who plan to undergo primary total knee arthroplasty on unilateral knee joint with a diagnosis of osteoarthritis or aseptic bone necrosis, but not of rheumatoid arthritis;
* All patients who have normal preoperative platelet count, normal prothrombin time, normal partial thromboplastin time, and normal international normalized ratio;
* The use of only balanced electrolyte solutions and/or albumin for plasma volume restitution

Exclusion Criteria:

* Allergy to tranexamic acid;
* Receiving warfarin or heparin; had a history of hemophilia, deep venous thrombosis, pulmonary embolism, or renal impairment; or were pregnant;
* Patients with any cardiovascular problems (such as myocardiac infarction history, atrial fibrillation, angina);
* Patients with thromboembolic disorders, or those exhibiting a deteriorating general condition;
* Preoperative anemia (a hemoglobin value of <11 g/dL in females and <12 g/dL in males), refusal of blood products;
* Preoperative use of anticoagulant therapy within five days before surgery, fibrinolytic disorders requiring intraoperative antifibrinolytic treatment, coagulopathy (as identified by a preoperative platelet count of <150,000/mm3, an international normalized ratio of >1.4, or a prolonged partial thromboplastin time [>1.4 times normal]).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Average amounts of transfusion | one week after surgery

SECONDARY OUTCOMES:
Calculated blood loss | one week after surgery
thrombosis | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China